CLINICAL TRIAL: NCT06671002
Title: Comparing Analgesic Regimen Effectiveness and Safety for Surgery for Kids (CARES for Kids) Trial
Brief Title: Comparing Analgesic Regimen Effectiveness and Safety for Surgery for Kids Trial
Acronym: CARES for Kids
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Mark Bicket, MD, PhD, Associate Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00252793; BPS-2023C1-32147 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Surgery; Pain, Post Operative
Keywords: Medications after surgery; NSAIDS; Acetaminophen; Opioids; Analgesics, non-narcotic; Tonsil removal; Gallbladder removal; Knee scope; Analgesics, opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Celecoxib; Analgesics, Opioid; Oxycodone; Hydromorphone; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Both study staff performing outcome assessment and data analysis will be masked to treatment assignment.
Who Masked: Outcomes Assessor
Masking Description: Both study staff performing outcome assessment and data analysis will be masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen/NSAID regimen (Other)
  Interventions: Drug: NSAID; Drug: Acetaminophen
- Acetaminophen/NSAID/Opioid regimen (Other)
  Interventions: Drug: Opioid; Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: NSAID — Once randomized to this group the surgical team will elect to prescribe 1 of the following treatment options for post-discharge pain:
  * Ibuprofen 10 milligrams(mg)/kilogram (kg) (maximum 600mg) by mouth every 6 hours around the clock for 2 days, then as needed for pain thereafter (40 doses)
  * Celecoxib 6mg/kg (maximum 400mg) by mouth once then 3 mg/kg (maximum 200mg) every 12 hours around the clock for 2 days, then as needed for pain thereafter (40 doses)
  Other Names: Ibuprofen; Celecoxib
  Arms: Acetaminophen/NSAID regimen
Drug: Opioid — Once randomized to this group the surgical team will elect to prescribe for 1 of the following treatment options to be given post procedure for post-discharge pain:
  * Oxycodone 0.1 mg/kg (maximum 5 mg) by mouth every 4 to 6 hours as needed for pain, number 10 doses.
  * Hydromorphone 0.04 mg/kg (maximum mg) by mouth 4 to 6 hours as needed, number 10 doses
  Other Names: Oxycodone; Hydromorphone
  Arms: Acetaminophen/NSAID/Opioid regimen
Drug: Acetaminophen — Participants will receive 15mg/kg up to 1000mg by mouth every 6 hours around the clock for the first 2 days after discharge from surgery then as needed thereafter (40 doses)
Drug: Ibuprofen — Ibuprofen 10mg/kg (maximum 600 mg) by mouth every 6 hours around the clock for 2 days after discharge from surgery then as needed thereafter (40 doses)
  Arms: Acetaminophen/NSAID/Opioid regimen

SUMMARY:
This trial is being completed to compare two commonly used options to treat pain after discharge from surgery. Participants that undergo tonsil removal, gallbladder removal, and knee scope will be eligible to enroll. Eligible participants will be randomized to prescription of 1 of 2 groups of medications (Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) plus acetaminophen or low dose opioids with the NSAIDs plus acetaminophen. The key question the study seeks to answer is which option will have the best outcomes and with the fewest side effects?

ELIGIBILITY:
Inclusion Criteria:

* No significant analgesic medication use before surgery as defined in the protocol
* Undergo one the following: elective tonsil removal (with or without adenoid removal), gallbladder removal (laparoscopic), and knee scope (arthroscopy).

Exclusion Criteria:

* Anticipated other surgery within 12 months
* Anticipated life expectancy of <12 months
* Those that have legal guardians (due to special permission to enroll in trials)
* Participants with complex chronic conditions per the Pediatric Medical Complexity Algorithm (e.g., trisomy 21)
* Patients with contraindications to non-steroidal anti-inflammatory drug (NSAID) drugs in the NSAID arm, opioid drugs in the opioid arm, or acetaminophen will be excluded.
* Liver disease
* Acute psychiatric instability (defined as current uncontrolled severe depression, severe post-traumatic stress disorder (PTSD), or suicidal ideation), substance use disorder not in remission or treatment, and history of diversion of controlled substances (opioids)

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness outcome - Pain intensity based on Brief Pain Inventory (BPI) pain intensity score at the surgical site over 14 days post-surgery | 14 days post-surgery, and up to 12 months after surgery
  This is a one question survey in which the worst pain intensity recorded (0-10 being the worst) will be used.
Safety outcome - number and severity of any adverse medication-related symptoms over 14 days post-surgery | 14 days post-surgery, and 1 month after surgery
  Symptom Checklist will proactively screen patients for reports of adverse events from analgesic medications over the first 14 days post-surgery.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Sleep Disturbance v1.0 short form 4a | Baseline and 1 month after surgery
  This is a 4-question survey in which participants will rate statements pertaining to quality of sleep. Participants will also rate sleep quality as very poor (5), poor (4), fair (3), good (2), or very good (1).
Patient Global Impression of Change (PGIC) | Day 7 up to 12 months after surgery
  The perception of improvement or worsening after treatment will be assessed by the patient global impression of change PGIC (range 0-7).
PROMIS Pediatric Pain Interference scale (Short form-8a) | Baseline up to 12 months after surgery
  This is an 8-question survey in which participants will rate statements pertaining to how pain interferes with activities and function.
Pain Catastrophizing Scale (PCS) | Baseline up to 12 months after surgery
  This is a 6-question survey in which participants will rate statements pertaining to their experience of pain.
Pediatric Quality of Life Inventory Short Form 15 | Baseline up to 12 months after surgery
  There are 15 questions with four scales for function related to physical, emotional, social, and school dimensions for adolescents. Participants answer questions from never (0) to almost always (4).
Quality of Recovery (QoR) 15 | Day 3, 1 week, and 2 weeks after surgery
  There are 15 questions assessed on a scale of 1-10, with 0 being none of the time and 10 being all of the time, 10 being the better outcome.
Patient Health Questionnaire (PHQ-2) | Baseline up to 12 months after surgery
  There are 2 questions that are completed to screen for depression. Participants answer from not at all (0) to Nearly every day (3). The scores range from 0-6 with a higher score indicating higher levels of depression.
Generalized Anxiety Disorder (GAD-2) | Baseline up to 12 months after surgery
  There are 2 questions that are completed to screen for anxiety. Participants answer from not at all (0) to Nearly every day (3). The scores range from 0-6 with a higher score indicating higher levels of anxiety.
Brief Screening Instrument for Adolescent Tobacco, Alcohol, and Drug Use | Baseline up to 12 months after surgery
  This is a 6-question survey about the participants' use of tobacco, alcohol and drugs.
National Survey on Drug Use and Health Questions on Opioid Misuse | Baseline up to 12 months after surgery
  This is a one question survey that assesses opioid misuse defined as use that is more than prescribed, for non pain-related reasons, or in a way not prescribed by a doctor.
New prolonged opioid use | Up to 12 months after surgery
  One question that will assess opioid prescription fills to identify new prolonged opioid use after surgery
Acute pain based on The Michigan Body Map | Up to 12 months after surgery
  Participants will document/mark on this image map to identify areas in which acute pain was felt.
Chronic pain based on Body Map | Up to 12 months after surgery
  Participants will document/mark on this image map to identify areas in which persistent or recurrent pain was felt.
Chronic pain based on Brief Pain Inventory (BPI) pain intensity score up to 12 months after surgery | to 12 months after surgery
  One question survey in which the participants rate pain intensity recorded (0-10), ten being the worst.
Healthcare Utilization related to pain | Up to 12 months after surgery
  Participants will answer questions about their healthcare utilization related to pain for the following three events: (1) postoperative clinical interactions related to pain in the form of patient messages, phone calls, and non-routine clinic visits related to pain, (2) emergency room visits, and (3) hospitalizations. The study team will also review health record for the same events.
Analgesic medication use | Up to 12 months after surgery
  Participants will answer questions about their analgesic medication use for acetaminophen, NSAIDs, opioids, and other medications, including prescription fills, over-the-counter use, and consumption. The study team will also review health record for prescription fills.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bicket, MD, PhD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles (CHLA), Los Angeles, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - University of Michigan, Ann Arbor, Michigan
  - Nationwide Children's (NCH), Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of the trial that is not subject to restrictions based on data sharing agreements (e.g., prescription drug monitoring program data), after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anticipated summer 2029 with no end date
Access Criteria: Investigators can access the IPD and supporting information for analyses related to aims in the proposal. The proposed used of the data needs to be approved by a review committee and the sponsor. Proposals may be submitted up to 36 months after data availability, after which data will be available in a data warehouse but without investigator support.

REFERENCES:
- See also: Project Summary on pcori.org — https://www.pcori.org/research-results/2023/comparing-two-ways-relieve-pain-after-surgery-among-youth-cares-kids-study